CLINICAL TRIAL: NCT06548100
Title: A Single-Arm, Open-Label, Safety Study in Patients With Generalized Lipodystrophy Switching From Metreleptin to Mibavademab, A Leptin Receptor Agonist Antibody
Brief Title: A Study of the Safety of Mibavademab in Pediatric and Adult Participants Switching From Metreleptin to Mibavademab for the Treatment of Generalized Lipodystrophy (GLD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R4461-GLD-2284; 2024-513202-54-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-07

CONDITIONS: Generalized Lipodystrophy
Keywords: Congenital or acquired generalized lipodystrophy; Leptin deficiency; Loss of subcutaneous tissue; Nutritional deprivation; Severe metabolic derangements; Severe diabetes mellitus; Hypertriglyceridemia; Berardinelli-Seip Syndrome; Lawrence Syndrome; Severe Insulin Resistance
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Obesity, Morbid; Diabetes Mellitus; Hypertriglyceridemia; Lipodystrophy, Familial Partial; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mibavademab (Experimental): Patients switching from at least 6 months of therapy with metreleptin to mibavademab.
  Interventions: Drug: mibavademab

INTERVENTIONS:
Drug: mibavademab — Administered by intravenous (IV) infusion followed by subcutaneous (SC) injection
  Other Names: REGN4461

SUMMARY:
This study is researching an experimental drug called mibavademab. The study is focused on participants with GLD who have been on metreleptin treatment for at least 6 months with no change in dose for the last 3 months.

The aim of the study is to see how safe and tolerable mibavademab is when switching from treatment with metreleptin.

The study is looking at several other research questions, including:

* What side effects may happen from taking mibavademab
* How much mibavademab is in the blood at different times
* Whether the body makes antibodies against mibavademab (which could make mibavademab less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of congenital or acquired GLD as defined by Multi-Society Practice Guidelines
2. Treatment with metreleptin for ≥6 months at time of screening at a stable dose, defined as no change in dose within the last 3 months prior to screening
3. Generally stable diet (based on participant's recall) and stable medication regimen for diabetes and/or dyslipidemia (in addition to metreleptin), for the last 3 months prior to screening
4. Willing and able to comply with clinic visits and study-related procedures. Participants who are unable/unwilling to self-inject, but are willing to have a capable caregiver inject, are considered eligible
5. Willing and able to provide, or have the treating physician provide, values of HbA1c and fasting triglycerides from at least 6 months prior to screening, as defined in the protocol

Key Exclusion Criteria:

1. Treatment with over-the-counter or prescription medications for weight loss within 3 months prior to the screening visit
2. Current chronic treatment with high-dose corticosteroids, as defined in the protocol
3. Any malignancy, eg, lymphoma, within the past 1 year, prior to screening visit except for fully treated basal cell or squamous epithelial cell carcinomas of the skin or carcinoma in situ of the cervix or anus
4. Estimated glomerular filtration rate (GFR) of <30 mL/min/1.73 m^2 based on chronic kidney disease epidemiology collaboration (CKD-EPI)/Schwartz equation at screening. Assessment can be repeated once
5. History of heart failure hospitalization, diagnosis of a myocardial infarction, stroke, clinically significant arrhythmia, transient ischemic attack, unstable angina, percutaneous or surgical revascularization procedure, or intracardiac device placement within 3 months before the screening visit, as defined in the protocol
6. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the participant by their participation in the study, as defined in the protocol

NOTE: Other protocol-defined inclusion / exclusion criteria apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to week 68
Severity of TEAEs | Up to week 68

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline, week 20 and week 52
Occurrence of HbA1c <7% | Week 20 and week 52
Occurrence of HbA1c <6.5% | Week 20 and week 52
Occurrence of requiring therapy with insulin in participants treated with mibavademab | Week 20 and week 52
Change in total insulin dose | Baseline, week 20 and week 52
Change in fasting plasma glucose | Baseline, week 20 and week 52
Percent change in fasting triglycerides | Baseline, week 20 and week 52
Occurrence of fasting triglycerides <500 mg/dL in participants treated with mibavademab | Baseline, week 20 and week 52
Occurrence of fasting triglycerides <200 mg/dL in participants treated with mibavademab | Baseline, week 20 and week 52
Occurrence of fasting triglycerides <150 mg/dL in participants treated with mibavademab | Baseline, week 20 and week 52
Concentrations of total mibavademab in serum | Up to week 68
Incidence of anti-drug antibodies (ADAs) to mibavademab | Up to week 68
Titer of ADAs to mibavademab | Up to week 68
Incidence of neutralizing antibodies (Nabs) to mibavademab | Up to week 68

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - National Institutes of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has :
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/